CLINICAL TRIAL: NCT03798769
Title: Supportive Oncology Care at Home for Patients With Pancreatic Cancer Receiving Preoperative FOLFIRINOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Ryan Nipp, Primary Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-532
Record Dates: First submitted 2018-12-27; First posted 2019-01-10 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Pancreas Cancer
Keywords: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Oncology Care at Home (Experimental): The Supportive Oncology Care at Home intervention entails the following:
  1. patient-reported symptoms, vital sign, and weight monitoring with appropriate triggers for phone calls and home visits by Medically Home based on a clinician-derived algorithm
  2. scheduled nursing visits for intravenous (IV) hydration during the course of chemotherapy;
  3. regular communication with oncology clinicians regarding care delivered at home to ensure continuity of care.
  Interventions: Other: Supportive Oncology Care at Home

INTERVENTIONS:
Other: Supportive Oncology Care at Home — Entails the following:
  1. patient-reported symptoms, vital sign, and weight monitoring with appropriate triggers to phone calls and home visits by Medically Home based on a clinician-derived algorithm;
  2. scheduled nursing visits for intravenous (IV) hydration during the course of chemotherapy;
  3. regular communication with oncology clinicians regarding care delivered at home to ensure continuity of care.

SUMMARY:
The goal of this research is to study an intervention, which the investigators call "Supportive Oncology Care at Home," that entails both remote patient monitoring (e.g. patient-reported symptoms, home monitored vital signs, and body weight) and a Medically Home care model (e.g. triggers for phone calls and visits to patients' homes to address and manage any concerning issues identified). Specifically, the investigators will conduct a single arm pilot study (N=20) in patients with pancreatic cancer who sign consent for parent trial of neoadjuvant FOLFIRINOX (18-179) receiving preoperative FOLFIRINOX to assess the feasibility and acceptability of Supportive Oncology Care at Home.

DETAILED DESCRIPTION:
Preoperative treatment can cause significant morbidity and often result in hospitalizations. Patients receiving preoperative FOLFIRINOX often experience numerous side effects, including nausea, vomiting, diarrhea, fatigue, fever, neuropathy, and loss of appetite. Frequently, patients require hospital admissions to help address uncontrolled symptoms related to their cancer and side effects related to the treatment,

Interventions targeting patients' symptoms and delivering care to patients at their homes have the potential to improve patient outcomes. Studies show that interventions targeting patients' symptoms can improve symptom management, enhance quality of life (QOL), and prevent hospitalizations.

Medically Home interventions have shown the potential to enhance patient outcomes. The Medically Home model of care is an alternative to a hospital admission for acute care and treatment of a clinical condition. Medically Home interventions entail providing medical care to acutely ill patients in their home. In addition, research in the general medicine literature has demonstrated that interventions involving remote patient monitoring with 'triggers' for visits to patients' homes for worrisome symptoms can enhance care outcomes.

Although this research demonstrates promising results, these studies have not been conducted among patients with cancer. Notably, the prior work involving home monitoring with visits as needed has lacked patient-reported outcomes, such as symptom monitoring. Thus, efforts are needed to develop and test interventions containing both symptom monitoring and the potential for home visits when necessary in a population of patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Within three weeks of signing consent for parent trial of neoadjuvant FOLFIRINOX
* Planning to receive care at Massachusetts General Hospital
* Ability to read and respond to questions in English
* Residing within 50 miles of Massachusetts General Hospital

Exclusion Criteria:

-Uncontrolled psychiatric illness or impaired cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Rates of study enrollment | 2 years
  Proportion of patients who agree to participate in the study and sign informed consent.
Rates of completion | 2 years
  Proportion of patients who complete daily patient-reported symptom assessments within the first two weeks of enrollment.

SECONDARY OUTCOMES:
Rates of completion of daily symptom monitoring | 2 years
  Proportion of participants completing daily symptom monitoring throughout the study
Rates of completion of daily vital signs | 2 years
  Proportion of participants completing daily reporting of vital signs throughout the study
Rates of completion of weekly body weight | 2 years
  Proportion of participants completing weekly reporting of body weight throughout the study
Number of home visits required | 2 years
  Number of home visits required, their average duration, the issues addressed at home, and the interventions delivered to patients at their home
Number of phone calls required | 2 years
  Number of phone calls required per patient as well as average duration of these calls
Number of emails required | 2 years
  Number of emails from Medically Home to the primary oncology team
Patient acceptability | 2 years
  Qualitative acceptability ratings from patients regarding helpfulness, convenience, and perceptions of the study.
Family caregiver acceptability | 2 years
  Qualitative acceptability ratings from family caregivers regarding helpfulness, convenience, and perceptions of the study.
Clinician acceptability | 2 years
  Qualitative acceptability ratings from clinicians regarding helpfulness, convenience, and perceptions of the study.
Number of emergency department visits | 2 Years
  The number of emergency department [ED] visits and the proportion of patients needing an emergency department [ED] visit
Number of urgent visits | 2 Years
  The number of urgent visits to clinic and the proportion of patients needing an urgent visit to clinic
Number of hospital admissions | 2 Years
  The number of hospital admissions and the proportion of patients needing a hospital admission
Change in symptom burden longitudinally throughout the study | 2 years
  Change in symptom burden (assessed using Edmonton Symptom Assessment System-revised [ESAS-r], range 0-10 for each symptom with higher scores indicating worse symptom burden) throughout the study.
Change in psychological distress | 2 years
  Change in psychological distress (assessed using the Patient Health Questionnaire-4 [PHQ-4], range 0-12 with higher scores indicating greater distress, and subscales for depression/anxiety ranging 0-6 with higher scores indicating greater distress) throughout the study.
Change in quality of life longitudinally throughout the study | 2 Years
  Change in quality of life (assessed using the Functional Assessment of Cancer Therapy-General [FACT-G], with range of 0-108 and higher scores indicating better quality of life) throughout the study.
Number of cycles of FOLFIRINOX received | 2 years
  Describe the number of cycles of FOLFIRINOX chemotherapy received by patients
Number of treatment delays | 2 years
  Describe the number of treatment delays for patients
Cumulative dose of FOLFIRINOX received | 2 years
  Describe the cumulative dose of FOLFIRINOX received

OTHER OUTCOMES:
Proportion of patients requiring a hospital admission | 2 years
  Compare difference in proportion of patients with hospital admissions between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Number of hospital admissions | 2 years
  Compare difference in number of hospital admissions between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of patients requiring an emergency department visit | 2 years
  Compare difference in proportion of patients with emergency department visits between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Number of emergency department visits | 2 years
  Compare difference in number of emergency department visits between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of patients requiring an urgent care visit | 2 years
  Compare difference in proportion of patients with urgent care visits between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Number of urgent care visits | 2 years
  Compare difference in number of urgent care visits between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of patients requiring a hospital admission or emergency department visit | 2 years
  Compare difference in proportion of patients with a hospital admission or emergency department visit between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Number of hospital admissions or emergency department visits | 2 years
  Compare difference in number of hospital admissions or emergency department visits between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of patients requiring a treatment delay | 2 years
  Compare difference in proportion of patients with a treatment delay between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of days in hospital or emergency department | 2 years
  Compare difference in proportion of days in hospital or emergency department between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Proportion of days in hospital, emergency department, or urgent care | 2 years
  Compare difference in proportion of days in hospital, emergency department, or urgent care between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Number of cycles of chemotherapy completed | 2 years
  Compare difference in number of cycles of chemotherapy completed between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Numbers of treatment delays | 2 years
  Compare difference in number of treatment delays between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Dose intensity | 2 years
  Compare difference in chemotherapy dose intensity between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Overall survival | 2 years
  Compare difference in overall survival between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home
Progression free survival | 2 years
  Compare difference in progression free survival between patients with pancreatic cancer receiving preoperative FOLFIRINOX who did and did not receive Supportive Oncology Care at Home

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Ryan Nipp, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor-Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor-Investigator or designee].

REFERENCES:
- [Derived] Nipp RD, Gaufberg E, Vyas C, Azoba C, Qian CL, Jaggers J, Weekes CD, Allen JN, Roeland EJ, Parikh AR, Miller L, Wo JY, Smith MH, Brown PMC, Shulman E, Fernandez-Del Castillo C, Kimmelman AC, Ting D, Hong TS, Greer JA, Ryan DP, Temel JS, El-Jawahri A. Supportive Oncology Care at Home Intervention for Patients With Pancreatic Cancer. JCO Oncol Pract. 2022 Oct;18(10):e1587-e1593. doi: 10.1200/OP.22.00088. Epub 2022 Jul 13. PMID 35830625